CLINICAL TRIAL: NCT00895336
Title: An Open Label Pilot Study of Lactobacillus GG in Pediatric Ulcerative Colitis
Brief Title: Lactobacillus GG in Pediatric Ulcerative Colitis (UC)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: IND for this study remained on clinical hold
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Lee Denson, M.D., Cincinnati Childrens
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0443
Record Dates: First submitted 2009-04-27; First posted 2009-05-08 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Ulcerative Colitis
Keywords: Pediatric Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative; Pediatric ulcerative colitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Lactobacillus GG — 1 capsule taken twice daily for a minimum of 28 days to a maximum of 35 days.
  Other Names: Culturelle

SUMMARY:
Abstract:

Current evidence suggests that the enteric flora is the primary trigger for chronic mucosal inflammation in the Inflammatory Bowel Diseases (IBD), Crohn's Disease (CD) and Ulcerative Colitis (UC). Studies using probiotic administration to modify the flora for either induction or maintenance of remission in IBD have had mixed results. Whether probiotics may exert an anti-inflammatory effect in IBD is not known. The investigators hypothesize that daily administration of a probiotic, Lactobacillus GG, for four weeks will reduce objective markers of mucosal inflammation in pediatric UC patients. The investigators will enroll 20 UC patients in remission or with mild disease activity. These patients will have a one month period of observation without intervention. They will then receive Lactobacillus GG (Culturelle), 1010 CFU by mouth twice a day for four weeks (28 days). At baseline and Day 28, and at day 56 clinical disease activity will be measured using the Pediatric UC Activity Index (PUCAI), a blood sample for determination of circulating granulocyte pSTAT3+ activation will be obtained, and a stool sample for determination of fecal calprotectin will be obtained. In addition, =the investigators will sample subject saliva to determine salivary glycan phenotype as a surrogate marker of changes of mucosal glycan expression in response to probiotic administration. The investigators anticipate that both circulating granulocyte pSTAT3+ activation and fecal calprotectin, as established biomarkers of colonic inflammation, will be reduced in subjects who receive Lactobacillus GG. Completion of the proposed studies will determine whether Lactobacillus GG reduces mucosal inflammation in pediatric UC, and will provide information to design a larger randomized trial.

The investigators' study design is novel in that it is the first probiotic study in children with UC and it will measure outcomes utilizing the biomarkers fecal calprotectin and pSTAT3+ circulating granulocytes.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent (and if applicable, Assent) and comply with study assessments for the full duration of the study;
* Enrolled without regard to gender, race, ethnicity;
* Age > 5 years to < 18 years;
* Diagnosis of Ulcerative Colitis (UC);
* Remission or mild disease activity defined by a PUCAI <34;
* Subjects taking stable doses (defined as 30 days) of all UC medications including AZA/6-MP, methotrexate, mesalamine, or infliximab at entry will be included;
* Willing to use birth control during study participation for females of child-bearing potential, as determined by investigator.

Exclusion Criteria:

* Current use, or use in the last 3 months, of probiotic preparations, not including yogurt;
* Known history of HIV or other known immunocompromised disease;
* Any central vascular line;
* Concomitant administration of an antibiotic, and must be off antibiotics for at least one month prior to enrollment;
* Cardiac valvular disease;
* Any other condition requiring current hospitalization for treatment;
* Current use of prednisone or budesonide;
* Diagnosis of Crohn's disease or indeterminate colitis;
* Pregnancy (positive pregnancy test) prior to enrollment in the study for females of child-bearing potential;
* Females of child-bearing potential who are unwilling to use birth control during study participation;
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated;
* Participation in another simultaneous clinical trial involving a drug or biological other than participation in the Pediatric IBD Registry and/or the Pediatric IBD Network for Research and Improvement.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be a reduction in the fecal calprotectin level following the receipt of study agent. | after dosing 28 - 35 days with LGG

CONTACTS AND LOCATIONS:
Overall Officials: Lee Denson, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States